CLINICAL TRIAL: NCT03747120
Title: Neoadjuvant Her2-targeted Therapy and Immunotherapy With Pembrolizumab (neoHIP)
Brief Title: Neoadjuvant Her2-targeted Therapy and Immunotherapy With Pembrolizumab [IIT2018-04-MCARTHUR-NEOHP]
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Heather McArthur, ASSOCIATE PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-0558
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: HER2-positive Breast Cancer; Breast Cancer
Keywords: her2-positive breast cancer; Breast Cancer; Pembrolizumab; Immunotherapy; Neoadjuvant her2 targeted therapy; Trastuzumab; Pertuzumab; Paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab; pertuzumab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: 1:1:1 randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: THP (Active Comparator): Arm A: Paclitaxel weekly x12 + Trastuzumab + Pertuzumab
  All subjects may receive standard of care systemic therapy after surgery per their treating physician's discretion.
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab
- Arm B: THP-Pembrolizumab (Experimental): Arm B: Paclitaxel weekly x12 + Trastuzumab + Pertuzumab + Pembrolizumab
  All subjects may receive standard of care systemic therapy after surgery per their treating physician's discretion.
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Pembrolizumab
- Arm C: TH-Pembrolizumab (Experimental): Arm C: Paclitaxel weekly x12 + Trastuzumab + Pembrolizumab
  All subjects may receive standard of care systemic therapy after surgery per their treating physician's discretion.
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Paclitaxel — All subjects will receive Paclitaxel weekly for 12 weeks
  Other Names: Taxol
Drug: Trastuzumab — All subjects will receive Trastuzumab every 3 weeks
  Other Names: Herceptin
Drug: Pertuzumab — Arm A and Arm B subjects will receive Pertuzumab every 3 weeks
  Other Names: Perjeta
  Arms: Arm A: THP; Arm B: THP-Pembrolizumab
Drug: Pembrolizumab — Arm B and Arm C subjects will receive Pembrolizumab every 3 weeks
  Other Names: Keytruda
  Arms: Arm B: THP-Pembrolizumab; Arm C: TH-Pembrolizumab

SUMMARY:
A phase 2 open-label, randomized, multi-center trial to evaluate the efficacy and safety of neoadjuvant trastuzumab, pertuzumab and weekly paclitaxel (THP) as compared to neoadjuvant trastuzumab, pertuzumab, pembrolizumab and weekly paclitaxel (THP-pembrolizumab), or neoadjuvant trastuzumab, pembrolizumab and weekly paclitaxel (TH-pembrolizumab ) in chemo naive patients with invasive human epidermal growth factor receptor 2 (HER2) positive breast cancer whose primary tumors are > 2 cm and/or clinically lymph node positive. Treatment will be followed by standard of care breast surgery and physician's choice adjuvant therapy per standard of care.

DETAILED DESCRIPTION:
A phase 2 open-label, randomized, multi-center trial to evaluate the efficacy and safety of neoadjuvant trastuzumab, pertuzumab and weekly paclitaxel (THP) as compared to neoadjuvant trastuzumab, pertuzumab, pembrolizumab and weekly paclitaxel (THP-pembrolizumab), or neoadjuvant trastuzumab, pembrolizumab and weekly paclitaxel (TH-pembrolizumab) in chemo naive patients with invasive human epidermal growth factor receptor 2 (HER2) positive breast cancer whose primary tumors are > 2 cm and/or clinically lymph node positive.

Patients will be randomized to either Arm A: THP (trastuzumab, pertuzumab and weekly paclitaxel), Arm B: THP-pembrolizumab (trastuzumab, pertuzumab, pembrolizumab) and weekly paclitaxel) or Arm C: TH-pembrolizumab (trastuzumab, pembrolizumab and weekly paclitaxel). Patients will be stratified according to hormone receptor status and lymph node status. All patients will be treated weekly every three weeks for four cycles (only paclitaxel will be administered weekly) and then undergo breast surgery. Arm A patients will be regarded as the reference group.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients with histologically confirmed invasive HER2-positive (by American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines) unilateral breast cancer
2. Have previously untreated non-metastaic (M0), cT2-4N0 or cT1-4N1-3 (biopsies of clinically suspicious lymph nodes to confirm nodal status is encouraged).
3. Multifocal/centric disease is permitted if all suspicious foci have been biopsied and are consistent with HER2-positive (by ASCO/CAP guidelines) invasive breast cancer
4. Be a male or female subject 18 years of age on the day of signing informed consent
5. Male Participants: A male participant must agree to use a contraception as detailed in Appendix C of this protocol during the treatment period and for at least 6 months after the last dose of study treatment and refrain from donating sperm during this period.
6. Female Participants: A female participant is eligible to participate if she is not pregnant (see Appendix C), not breastfeeding, and at least one of the following conditions applies: a.) Not a woman of childbearing potential (WOCBP) as defined in Appendix C OR b.) A WOCBP who agrees to follow the contraceptive guidance in Appendix C during the treatment period and for at least 6 months after the last dose of study treatment.
7. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
8. Provides adequate archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue. Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
10. Have adequate organ function as defined by the following parameters. Specimens must be collected within 7 days prior to the start of study treatment.

    * Absolute neutrophil count (ANC) ≥1500/µL
    * Platelets ≥100 000/µL
    * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La
    * Renal Creatinine (≤1.5 × ULN OR) OR Measured or calculated(b) creatinine clearance (≥30 mL/min for participant with creatinine levels) (GFR can also be used in place of creatinine or CrCl) (>1.5 × institutional ULN)
    * Hepatic Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN aspartate aminotransferase (AST, SGOT) and alanine aminotransferase (ALT, SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
    * Coagulation International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
    * Cardiac Echocardiogram or MUGA (multigated radionuclide angiography) Baseline LVEF ≥ 55%

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
2. Has received prior therapy with an anti-PD-1 (programmed death protein 1), anti-PD-L1 (Programmed death-ligand 1), or anti PD L2 (Programmed death-ligand 2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to randomization. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active systemic treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a known history of Human Immunodeficiency Virus (HIV).
13. Has a known active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C virus (i.d. HCV RNA [qualitative] is detected) infection.
14. Has a known history of active TB (Bacillus Tuberculosis).
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
18. Has significant cardiovascular disease, such as:

    * History of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months
    * Congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA class III or IV
    * Angina pectoris requiring anti-anginal medication, uncontrolled arrhythmias, or uncontrolled hypertension (systolic blood pressure > 180mmHg and/or diastolic blood pressure > 100mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2029-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Heather McArthur, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (5):
- United States (5):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Providence Cancer Institute, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: THP: Arm A: Paclitaxel weekly x12 + Trastuzumab + Pertuzumab
  All subjects may receive standard of care systemic therapy after surgery per their treating physician's discretion.
  Paclitaxel: All subjects will receive Paclitaxel weekly for 12 weeks
  Trastuzumab: All subjects will receive Trastuzumab every 3 weeks
  Pertuzumab: Arm A and Arm B subjects will receive Pertuzumab every 3 weeks
- Arm B: THP-Pembrolizumab: Arm B: Paclitaxel weekly x12 + Trastuzumab + Pertuzumab + Pembrolizumab
  All subjects may receive standard of care systemic therapy after surgery per their treating physician's discretion.
  Paclitaxel: All subjects will receive Paclitaxel weekly for 12 weeks
  Trastuzumab: All subjects will receive Trastuzumab every 3 weeks
  Pertuzumab: Arm A and Arm B subjects will receive Pertuzumab every 3 weeks
  Pembrolizumab: Arm B and Arm C subjects will receive Pembrolizumab every 3 weeks
- Arm C: TH-Pembrolizumab: Arm C: Paclitaxel weekly x12 + Trastuzumab + Pembrolizumab
  All subjects may receive standard of care systemic therapy after surgery per their treating physician's discretion.
  Paclitaxel: All subjects will receive Paclitaxel weekly for 12 weeks
  Trastuzumab: All subjects will receive Trastuzumab every 3 weeks
  Pembrolizumab: Arm B and Arm C subjects will receive Pembrolizumab every 3 weeks
Period: Overall Study
Arm/Group | Arm A: THP | Arm B: THP-Pembrolizumab | Arm C: TH-Pembrolizumab
Started | 58 | 58 | 22
Completed | 55 | 57 | 20
Not Completed | 3 | 1 | 2
Not completed — treatment related toxicity | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: THP | Arm B: THP-Pembrolizumab | Arm C: TH-Pembrolizumab | Total
Number analyzed (Participants) | 58 | 58 | 22 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 49 | 19 | 113
  >=65 years | 13 | 9 | 3 | 25
Age, Continuous [Mean (Full Range); unit: years] | 53.52 [32 to 79] | 52.24 [28 to 82] | 51.59 [32 to 74] | 52.67 [28 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 22 | 137
  Male | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 12 | 1 | 27
  Not Hispanic or Latino | 44 | 46 | 21 | 111
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 7 | 6 | 2 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 0 | 6
  White | 46 | 47 | 20 | 113
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 58 | 58 | 22 | 138

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR)
Description: Proportion of subjects without residual invasive cancer in the breast and axilla from randomization to definitive surgery.
  - Residual invasive cancer defined based on hematoxylin and eosin evaluation of complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by pathologist assessment.
Time Frame: 16 weeks from randomization
Population: Data shown are for the intention-to-treat population, which is defined as any subject who was randomized regardless of treatment completion. Participants were classified as non-responders if they did not receive study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: THP | Arm B: THP-Pembrolizumab | Arm C: TH-Pembrolizumab
Number analyzed (Participants) | 58 | 58 | 22
Participants | 28 | 39 | 5

2. Secondary Outcome: Pathological Complete Invasive and in Situ Response Rate (Breast and Axilla)
Description: Proportion of subjects without residual invasive and in situ cancer in the breast and axilla disease from randomization to definitive surgery.
  - Residual invasive cancer and in situ disease defined based on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by pathological assessment.
Time Frame: 16 weeks from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: THP | Arm B: THP-Pembrolizumab | Arm C: TH-Pembrolizumab
Number analyzed (Participants) | 58 | 58 | 22
Participants | 25 | 30 | 4

3. Secondary Outcome: Pathological Complete Response Rate (pCR) in Breast Only
Description: Proportion of subjects without residual invasive cancer in the breast from randomization to definitive surgery.
  - Residual invasive breast cancer defined based on hematoxylin and eosin evaluation of the complete resected breast specimen following completion of neoadjuvant systemic therapy by pathological assessment.
Time Frame: 16 weeks from randomization
Population: Data shown are for the intention-to-treat population, which is defined as any subject who was randomized regardless of treatment completion. Participants were classified as non-responders if they did not receive study medication or had missing data regarding pathological complete response for any reason.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: THP | Arm B: THP-Pembrolizumab | Arm C: TH-Pembrolizumab
Number analyzed (Participants) | 58 | 58 | 22
Participants | 28 | 39 | 5

4. Secondary Outcome: Residual Cancer Burden (RCB)
Description: Proportion of subjects with RCB 0-I, II or III from randomization to definitive surgery.
  -Residual Cancer Burden defined based on the RCB index, a component of four pathological parameters: bi-dimensional diameter of primary tumor bed, percent of cellularity in the tumor bed, number of involved lymph nodes and size of the largest nodal metastasis.
  The RCB possible scores are:
  * RCB-0: Represents a pathologic complete response (pCR), meaning no residual invasive breast cancer was found after neoadjuvant therapy.
  * RCB-I: Indicates a minimal residual disease burden.
  * RCB-II: Represents a moderate residual disease burden.
  * RCB-III: Indicates an extensive residual disease burden. Therefore, higher score indicates worse outcome.
Time Frame: 16 weeks from randomization
Population: RCB was evaluated among the modified intention-to-treat population, defined as patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: THP | Arm B: THP-Pembrolizumab | Arm C: TH-Pembrolizumab
Number analyzed (Participants) | 58 | 58 | 20
Participants
  RBC-0-1 | 39 | 44 | 13
  RBC-2 | 14 | 12 | 6
  RBC-3 | 5 | 2 | 1

5. Secondary Outcome: Breast Conserving Surgery Rate
Description: Proportion of subjects who achieved breast conserving surgery out of the intent-to-treat population without inflammatory breast cancer from randomization to definitive surgery (breast conserving surgery).
Time Frame: 16 weeks from randomization
Reporting Status: Not Posted

6. Secondary Outcome: Event Free Survival
Description: Mean difference in time (in months) from randomization to any of the following events progression of disease that precludes surgery, local or distant recurrence, or death due to any cause.
Time Frame: 36 months from randomization
Reporting Status: Not Posted

7. Secondary Outcome: Invasive Disease-free Survival (IDFS)
Description: Mean difference in time (in months) from date of surgery (date of no disease) to the first documentation of invasive progressive disease or death.
Time Frame: 33 months from surgery
Reporting Status: Not Posted

8. Secondary Outcome: Overall Survival
Description: Mean difference in time (in months) from randomization to death.
Time Frame: 36 months from randomization
Reporting Status: Not Posted

9. Secondary Outcome: Symptomatic Cardiac Events and Asymptomatic LVEF Events
Description: This outcome measure was inadvertently included in the original registration of the record (by a different organization- this is a transfer record). This specific outcome was never a pre-specified outcome within any version of the protocol. The error was not caught until we began to enter and report results. No data was ever collected for this outcome and hence no data can be reported. There is no plan to collect or analyze data in the future as the outcome was added in error and should have been removed prior to reporting results.
Time Frame: 36 months from randomization
Population: This outcome measure was inadvertently added at the time of registration but since it is not a pre-specified outcome within the protocol, no data was collected for this outcome and hence no data to report here.
Arm/Group | Arm A: THP | Arm B: THP-Pembrolizumab | Arm C: TH-Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: AEs and SAEs
Description: Incidence and severity of adverse events (AE) and serious adverse events (SAE) from cycle 1 day 1 until 30 days post-surgery.
  -AEs and SAEs based on CTCAE 5.0
Time Frame: 20 weeks from treatment initiation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Averse event data were collected during the neoadjuvant phase, which spans from the initiation of treatment to the day of surgery, 16 weeks.
Description: 22 patients were randomized to Arm C; however, two patients withdrew consent before study treatment was initiated. SAE/AE analysis was conducted in the safety population which is defined as patients who had a least one dose of study treatment.
Arm/Group | Arm A: THP | Arm B: THP-Pembrolizumab | Arm C: TH-Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/58 | 3/58 | 1/20
Other Adverse Events (participants affected / at risk) | 39/58 | 33/58 | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: THP (N=58) | Arm B: THP-Pembrolizumab (N=58) | Arm C: TH-Pembrolizumab (N=20)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: THP (N=58) | Arm B: THP-Pembrolizumab (N=58) | Arm C: TH-Pembrolizumab (N=20)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (14) | 13 (16) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 15 (23) | 10 (23) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 24 (34) | 26 (38) | 3 (3)
Elevated ALT (Hepatobiliary disorders) | 10 (18) | 7 (13) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 13 (14) | 3 (3)
Fatigue (General disorders) | 21 (25) | 19 (22) | 3 (4)
Headache (Nervous system disorders) | 10 (13) | 7 (7) | 2 (2)
Insomnia (Psychiatric disorders) | 11 (12) | 5 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 18 (22) | 15 (21) | 4 (4)
Peripheral Neuropathy (Nervous system disorders) | 15 (18) | 13 (20) | 5 (12)
Rash (Skin and subcutaneous tissue disorders) | 12 (18) | 19 (48) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (7) | 6 (9) | 4 (6)
Vomitting (Gastrointestinal disorders) | 5 (8) | 4 (6) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT03747120/Prot_SAP_000.pdf